CLINICAL TRIAL: NCT02000310
Title: Investigation of Molecular and Cellular Mechanisms of Lysosomal Storage Diseases
Brief Title: Molecular and Cellular Mechanisms of Lysosomal Storage Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: O & O Alpan LLC (Other)
Responsible Party: Sponsor
Other Study IDs: 13-CFCT-07
Record Dates: First submitted 2013-11-25; First posted 2013-12-04 (Estimated); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Lysosomal Storage Disorders
Keywords: Gaucher disease; Fabry disease; Pompe disease; Niemann-Pick disease
MeSH Terms: conditions — Lysosomal Storage Diseases; Gaucher Disease; Fabry Disease; Glycogen Storage Disease Type II; Niemann-Pick Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The lysosome is a specialized part of the cell that functions to degrade metabolic wastes in the cell. Defects in the functioning of the lysosome result in accumulation and subsequent storage of such metabolic wastes. These defects lead to conditions known as lysosomal storage diseases (LSD). LSDs are caused by inherited genetic mutations and there are over 40 genetically distinct lysosomal storage diseases. Within each specific lysosomal storage disease there are variances in severity of disease, age of onset, and clinical presentation. Though the genetic mutations contributing to the disease have been largely clarified, the molecular and cellular mechanisms that contribute to variations in each distinct LSD remain unclear. With this study we intend to better understand at the cellular and molecular level how the accumulation and storage of metabolic wastes in the lysosome affect the clinical manifestation of LSDs, to detect changes in these mechanisms upon treatment administration, and to correlate these results to genetic information. The knowledge obtained from this research study could lead to better ways to diagnose and treat lysosomal storage diseases.

ELIGIBILITY:
Inclusion Criteria:

* Subject is greater than or equal to 1 day of age and less than or equal to 100 years of age
* Signed Informed Consent/Assent
* Subject is able and willing to comply with study protocol requirements.
* From clinical or blood laboratory findings subject has evidence of a lysosomal storage disease or a family member of a patient with lysosomal storage disease

Exclusion Criteria:

* Pregnant woman

Ages: 1 Day to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients or suspected carriers of a lysosomal storage disorders.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2013-11 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Correlating genetic mutations with clinical signs and symptoms | 5 years
  Genetic information (DNA) will be collected from biological samples (e.g. blood, skin cells) and correlated with clinical signs and symptoms. DNA will be sequenced in order to identify a specific mutation. Fluorescence assay will be performed to measure the enzyme activity of the affected protein. Physical examination will be performed, and supporting test results will be collected for identifying the signs and symptoms of the particular disorder.

SECONDARY OUTCOMES:
Associated Immune Pathophysiology | 5 years
  Blood will be collected for identifying alterations in the innate and adaptive immune system. Flow cytometry will be used to analyze cell surface and intracellular biomarkers on immune cells such as B-cells, T-cells, eosinophils.

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Goker-Alpan, MD, Principal Investigator — Lysosomal & Rare Disorders Research & Treatment Center (LDRTC); Renuka Limgala, PhD, Principal Investigator — LDRTC
Locations (1):
- Lysosomal and Rare Disorders Research and Treatment Center, Inc (LDRTC), Fairfax, Virginia, United States